CLINICAL TRIAL: NCT00281268
Title: Fluids and Catheters Treatment Trial (FACTT) - ARDS Clinical Research Network
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: ARDSNet (Other)
Model: Factorial | Purpose: Treatment
Other Study IDs: 356
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2008-01-21 (Estimated); Status verified 2008-01

CONDITIONS: Acute Respiratory Distress Syndrome; Lung Diseases
MeSH Terms: conditions — Respiratory Distress Syndrome; Lung Diseases | interventions — Central Venous Catheters

INTERVENTIONS:
Procedure: pulmonary artery catheter
Procedure: central venous catheter
Procedure: fluid management

SUMMARY:
To assess rapidly innovative treatment methods in patients with adult respiratory distress syndrome as well as those at risk of developing ARDS.

DETAILED DESCRIPTION:
BACKGROUND:

Adult respiratory distress syndrome affects approximately 150,000 people in the United States each year. Despite twenty years of research into the mechanisms that cause this syndrome and numerous developments in the technology of mechanical ventilation, the mortality has remained greater than 50 percent. Many of the patients are young, and in addition to the tragic loss of human life, can be added the cost to society because these patients spend an average of two weeks in intensive care units and require multiple high tech procedures. Because of the overwhelming nature of the lung injury once it is established, prevention would appear to be the most effective strategy for improving the outlook in this condition.

Basic research has identified numerous inflammatory pathways that are associated with the development of ARDS. Agents that block these mediators prolong survival in animals with lung injury, and a few of them have been tested in patients. Because of the large number of putative mediators and the variety of ways that their action can be blocked, the possibility for new drug development is almost infinite. This is an exciting prospect, since it envisions the first effective pharmacologic treatment for ARDS. However, preliminary clinical studies have shown conflicting results, and there is an urgent need for a mechanism to efficiently and effectively test new drugs in ARDS.

Treatment studies in patients with ARDS are difficult to perform for three reasons. The complicated clinical picture makes it difficult to accumulate a large number of comparable patients in any one center. There is no agreement on the optimal supportive care of these critically ill patients. Many of the patients meeting study criteria will not be enrolled in study protocols because of the acute nature of the disease process. For these reasons, therapeutic trials in ARDS require multicenter cooperation.

DESIGN NARRATIVE:

Network investigators have developed a plan for a new protocol to assess the Pulmonary Artery Catheter as a management tool in ARDS. The new study was prompted by recommendations from the FDA/NIH Pulmonary Artery Catheter Clinical Outcomes workshop convened in August 1997 in response to concerns in the medical community regarding the clinical benefit and safety of pulmonary artery catheters. The new protocol in the Fluids and Catheters Treatment Trial (FACTT) is a two by two factorial design comparing the patients receiving PAC or a central venous catheter (CVC) with one of two fluid management strategies (conservative vs. liberal). The randomized, multicenter trial is designed to include 1000 patients. The primary endpoint is mortality at 60 days. Secondary endpoints include ventilator free days and organ failure free days.

ELIGIBILITY:
Men and women, 13 years of age or older, with ARDS or risk factors for ARDS. Patients will be considered at risk if they are critically ill and have trauma, sepsis, shock, pneumonia, inhalation injury, drug overdose, pancreatitis, hypertransfusion.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Abraham — University of Colorado, Denver; Antonio Anzueto — University of Texas; Alfred Connors — University of Virginia; Bennett deBoisblanc — Louisiana State University Health Sciences Center in New Orleans; Michael Donahoe — University of Pittsburgh; William Fulkerson — Duke University; Kalpalatha Guntupalli — Baylor College of Medicine; Robert Hite — Wake Forest University; Leonard Hudson — University of Washington; Paul Lanken — University of Pennsylvania; Michael Matthay — University of California; Alan Morris — Latter Day Saints Hospital; James Russell — University of British Columbia; Gregory Schmidt — University of Chicago; David Schoenfeld — Massachusetts General Hospital; Henry Silverman — University of Maryland; Jay Steingrub — Baystate Medical Center; Galen Toews — University of Michigan; Arthur Wheeler — Vanderbilt University; Herbert Wiedemann — The Cleveland Clinic

REFERENCES:
- [Derived] Bhatraju P, Hsu C, Mukherjee P, Glavan BJ, Burt A, Mikacenic C, Himmelfarb J, Wurfel M. Associations between single nucleotide polymorphisms in the FAS pathway and acute kidney injury. Crit Care. 2015 Oct 19;19:368. doi: 10.1186/s13054-015-1084-5. PMID 26477820
- [Derived] Stewart RM, Park PK, Hunt JP, McIntyre RC Jr, McCarthy J, Zarzabal LA, Michalek JE; National Institutes of Health/National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome Clinical Trials Network. Less is more: improved outcomes in surgical patients with conservative fluid administration and central venous catheter monitoring. J Am Coll Surg. 2009 May;208(5):725-35; discussion 735-7. doi: 10.1016/j.jamcollsurg.2009.01.026. Epub 2009 Mar 31. PMID 19476825
- [Derived] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wheeler AP, Bernard GR, Thompson BT, Schoenfeld D, Wiedemann HP, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Pulmonary-artery versus central venous catheter to guide treatment of acute lung injury. N Engl J Med. 2006 May 25;354(21):2213-24. doi: 10.1056/NEJMoa061895. Epub 2006 May 21. PMID 16714768
- [Derived] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wiedemann HP, Wheeler AP, Bernard GR, Thompson BT, Hayden D, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Comparison of two fluid-management strategies in acute lung injury. N Engl J Med. 2006 Jun 15;354(24):2564-75. doi: 10.1056/NEJMoa062200. Epub 2006 May 21. PMID 16714767
- See also: Acute Respiratory Distress Syndrome Clinical Network (ARDSNet) — http://www.ardsnet.org